CLINICAL TRIAL: NCT01996436
Title: The Intra-arterial Vasospasm Trial - A Multi-center Randomized Study
Brief Title: The Intra-arterial Vasospasm Trial
Acronym: iVAST
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Peng Roc Chen, MD (Other)
Collaborators: Yale University (Other); Thomas Jefferson University (Other); University of Illinois at Chicago (Other); Wake Forest University Health Sciences (Other); Temple University (Other); Geisinger Clinic (Other); Northwell Health (Other); University of Michigan (Other); Lenox Hill Hospital (Other); Weatherhead Foundation (Unknown); University of California, Irvine (Other)
Responsible Party: Sponsor-Investigator, Peng Roc Chen, MD, Professor in Neurosurgery, The University of Texas Health Science Center, Houston
Organization: The University of Texas Health Science Center, Houston (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IVT_201310 (HSC-MS-13-0586)
Record Dates: First submitted 2013-11-12; First posted 2013-11-27 (Estimated); Results first posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Vasospasm
Keywords: cerebral vasospasm; aneurysmal subarachnoid hemorrhage; intra arterial drug treatment for cerebral vasospasm; nicardipine milrinone nitroglycerin verapamil
MeSH Terms: conditions — Vasospasm, Intracranial; Subarachnoid Hemorrhage | interventions — Nicardipine; Verapamil; Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Nicardipine (Active Comparator): Group 1 : Nicardipine 5mg per circulation intra-arterial injection, Pharmacological angioplasty
  Interventions: Drug: Nicardipine
- Verapamil (Active Comparator): Group 3: Verapamil 10mg per circulation intra-arterial injection, Pharmacological angioplasty
  Interventions: Drug: Verapamil
- Nicardipine + Verapamil + Nitroglycerin (Active Comparator): Group 4 : Nicardipine 5mg + Verapamil 10mg + Nitroglycerin 200mcg in 4cc 5 % dextrose in water , intra-arterial injection, Pharmacological angioplasty
  Interventions: Drug: Nicardipine + Verapamil + Nitroglycerin

INTERVENTIONS:
Drug: Nicardipine — Pharmacological angioplasty: intra-arterial drug infusion via catheter to treat cerebral vasospasm
  Other Names: Cardene
  Arms: Nicardipine
Drug: Verapamil — Pharmacological angioplasty: intra-arterial drug infusion via catheter to treat cerebral vasospasm
  Arms: Verapamil
Drug: Nicardipine + Verapamil + Nitroglycerin — Pharmacological angioplasty: intra-arterial drug infusion via catheter to treat cerebral vasospasm
  Arms: Nicardipine + Verapamil + Nitroglycerin

SUMMARY:
The primary objective of the study is to determine the optimal intra-arterial drug treatment regimen for arterial lumen restoration post cerebral vasospasm following aneurysmal subarachnoid hemorrhage. The secondary objective is to evaluate clinical outcome at 90 days post discharge following optimal intra-arterial drug treatment for cerebral vasospasm.

We hypothesize that Intra-arterial (IA) infusion of a combination of multiple vasodilators is more efficacious than single agent treatment cerebral vasospasm therapy.

All procedures done as a part of this study are standard hospital care procedures done to treat cerebral vasospasm and all drugs to be used are FDA approved.

DETAILED DESCRIPTION:
The primary objective of the study is to determine the optimal intra-arterial drug treatment regimen for arterial lumen restoration post cerebral vasospasm following aneurysmal subarachnoid hemorrhage.

The secondary objective is to evaluate clinical outcome at 90 days post discharge following optimal intra-arterial drug treatment for cerebral vasospasm.

This study is a prospective multicenter randomized trial. The primary outcome measure is the Post infusion improvement ratio (PIIR) assessed 10 minutes after completion of the intra-arterial infusion. PIIR is a measure of arterial lumen diameter pre and post intra-arterial drug infusion in the presenting vasospasmic blood vessel.

Modified Rankin score (mRS) at 3 months post hospital discharge will be recorded as a secondary outcome to assess clinical outcome.

The interventions in this study are a part of routine standard of care (SOC) procedures for cerebral vasospasm treatment. Following surgical or endovascular intervention for aneurysmal Subarachnoid Hemorrhage (aSAH) if patients develop cerebral vasospasm refractory to maximal medical management, endovascular treatment by intra-arterial drug infusion of single drug agent or cocktail drug agents will be initiated.

Study participants will be randomly assigned to one of the three treatment groups where one single drug agent or cocktail drug agents will be intra-arterially administered. Pre & post infusion vasospasmic vessel diameters will be compared. The change in diameter will be quantified based on the mean percentage change. Three months post hospital discharge, study participants will be followed up in clinic to evaluate clinical outcome.

The study will require 330 patients in total. The patient population will be hospitalized patients presenting with cerebral vasospasm post aneurysmal subarachnoid hemorrhage.

Subjects will be stratified by randomization into 3 treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, age 18-80 years old, with ruptured aneurysm(s) who experience cerebral vasospasm post operatively within 3-21 days.
* Symptomatic vasospasm (clinical or TCD)
* For centers that perform a routine day 7 angiogram post-aneurysm treatment - 50% or more stenosis seen on diagnostic angiogram for asymptomatic patients.

Exclusion Criteria:

* Inability to obtain consent from patient or patients kin
* Pregnant women
* less than 18 years of age of more than 80 years of age
* Hunt Hess Grade 5 SAH
* Intra-arterial drug treatment in all 3 arterial territories

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peng R Chen, MD, Principal Investigator — University of Texas Medical School at Houston; Ketan R Bulsara, MD, MBA, Principal Investigator — UConn Health
Locations (5):
- United States (5):
  - Yale School of Medicine, New Haven, Connecticut
  - Northwell Health, Manhasset, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Geisinger Clinic, Danville, Pennsylvania
  - University of Texas Medical School at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dorsch NW, King MT. A review of cerebral vasospasm in aneurysmal subarachnoid haemorrhage Part I: Incidence and effects. J Clin Neurosci. 1994 Jan;1(1):19-26. doi: 10.1016/0967-5868(94)90005-1. PMID 18638721
- [Background] Treggiari MM, Walder B, Suter PM, Romand JA. Systematic review of the prevention of delayed ischemic neurological deficits with hypertension, hypervolemia, and hemodilution therapy following subarachnoid hemorrhage. J Neurosurg. 2003 May;98(5):978-84. doi: 10.3171/jns.2003.98.5.0978. PMID 12744357
- [Background] Biller J, Godersky JC, Adams HP Jr. Management of aneurysmal subarachnoid hemorrhage. Stroke. 1988 Oct;19(10):1300-5. doi: 10.1161/01.str.19.10.1300. No abstract available. PMID 3176090
- [Background] Kassell NF, Sasaki T, Colohan AR, Nazar G. Cerebral vasospasm following aneurysmal subarachnoid hemorrhage. Stroke. 1985 Jul-Aug;16(4):562-72. doi: 10.1161/01.str.16.4.562. PMID 3895589
- [Background] Keuskamp J, Murali R, Chao KH. High-dose intraarterial verapamil in the treatment of cerebral vasospasm after aneurysmal subarachnoid hemorrhage. J Neurosurg. 2008 Mar;108(3):458-63. doi: 10.3171/JNS/2008/108/3/0458. PMID 18312091
- [Background] Linfante I, Delgado-Mederos R, Andreone V, Gounis M, Hendricks L, Wakhloo AK. Angiographic and hemodynamic effect of high concentration of intra-arterial nicardipine in cerebral vasospasm. Neurosurgery. 2008 Dec;63(6):1080-6; discussion 1086-7. doi: 10.1227/01.NEU.0000327698.66596.35. PMID 19057319
- [Background] Badjatia N, Topcuoglu MA, Pryor JC, Rabinov JD, Ogilvy CS, Carter BS, Rordorf GA. Preliminary experience with intra-arterial nicardipine as a treatment for cerebral vasospasm. AJNR Am J Neuroradiol. 2004 May;25(5):819-26. PMID 15140728
- [Background] Pierot L, Aggour M, Moret J. Vasospasm after aneurysmal subarachnoid hemorrhage: recent advances in endovascular management. Curr Opin Crit Care. 2010 Apr;16(2):110-6. doi: 10.1097/MCC.0b013e3283372ef2. PMID 20098322
- [Background] Fraticelli AT, Cholley BP, Losser MR, Saint Maurice JP, Payen D. Milrinone for the treatment of cerebral vasospasm after aneurysmal subarachnoid hemorrhage. Stroke. 2008 Mar;39(3):893-8. doi: 10.1161/STROKEAHA.107.492447. Epub 2008 Jan 31. PMID 18239182

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 92 enrolled participants, 91 met inclusion criteria and were randomized to treatment.
Period: Overall Study
Arm/Group | Nicardipine | Verapamil | Nicardipine + Verapamil + Nitroglycerin
Started | 32 | 31 | 29
Received Intervention | 32 | 30 | 29
Completed | 32 | 30 | 29
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Includes all participants who received intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicardipine | Verapamil | Nicardipine + Verapamil + Nitroglycerin | Total
Number analyzed (Participants) | 32 | 30 | 29 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (13.081) | 50.933 (13.769) | 50.482 (10.796) | 51.164 (12.652)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 21 | 18 | 63
  Male | 8 | 9 | 11 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 5 | 19
  Not Hispanic or Latino | 19 | 18 | 21 | 58
  Unknown or Not Reported | 6 | 5 | 3 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 8 | 5 | 16
  White | 15 | 9 | 14 | 38
  More than one race | 2 | 2 | 1 | 5
  Unknown or Not Reported | 10 | 9 | 9 | 28
Region of Enrollment [Number; unit: participants]
  United States | 32 | 30 | 29 | 92
Weight [Mean (Standard Deviation); unit: pounds (lbs)] | 185.082 (50.179) | 166.402 (39.156) | 193.338 (45.524) | 181.554 (45.295)
Height [Mean (Standard Deviation); unit: centimeters] | 161.667 (19.527) | 167.674 (8.741) | 169.889 (8.801) | 166.267 (13.570)
Number of Participants with history of hypertension [Count of Participants; unit: Participants] | 17 | 17 | 18 | 52
Number of Participants with history of diabetes mellitus 1 or 2 [Count of Participants; unit: Participants] | 6 | 4 | 6 | 16
Number of participants with morbid obesity [Count of Participants; unit: Participants] | 6 | 4 | 2 | 12
Smoking History [Count of Participants; unit: Participants]
  Current Smoker | 11 | 9 | 12 | 32
  Non-Smoker | 14 | 16 | 11 | 41
  Past Smoker | 3 | 2 | 4 | 9
  Unknown | 4 | 3 | 2 | 9
Alcohol History [Count of Participants; unit: Participants]
  Habitual Alcoholic | 2 | 3 | 2 | 7
  Social Drinker | 7 | 10 | 8 | 25
  Teetotaler | 12 | 10 | 12 | 34
  Unknown | 11 | 7 | 7 | 25
Substance Abuse History [Count of Participants; unit: Participants]
  Cocaine | 3 | 0 | 2 | 5
  Heroin | 0 | 0 | 0 | 0
  Crystal Meth | 0 | 0 | 0 | 0
  Cannabis | 2 | 2 | 4 | 8
  Prescription Drugs | 0 | 2 | 0 | 2
  No Substance abuse | 21 | 19 | 19 | 59
  Unknown | 7 | 9 | 6 | 22
Number of Participants with History of Hypercholesterolemia [Count of Participants; unit: Participants] | 6 | 5 | 3 | 14

OUTCOME MEASURES:

1. Primary Outcome: Post Infusion Improvement Ratio (PIIR)
Description: Post infusion improvement ratio (PIIR) = ((B - A) / A) *100
  A = pre-infusion blood vessel diameter B = post infusion blood vessel diameter
Time Frame: pre pharmacological angioplasty blood vessel diameter - 0 min, post pharmacological angioplasty blood vessel diameter- 10 min after infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Nicardipine | Verapamil | Nicardipine + Verapamil + Nitroglycerin
Number analyzed (Participants) | 18 | 24 | 17
Participants
  Below 30% | 4 | 3 | 2
  30% to 50% | 10 | 14 | 8
  51% to 70% | 1 | 6 | 5
  Above 70% | 3 | 1 | 2

2. Secondary Outcome: Disability or Dependence in Daily Activities as Assessed by the Modified Rankin Score
Description: The modified Rankin Scale (mRS) is used to assess the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.
  The Modified Rankin Score (mRS) is scored as follows:
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
Time Frame: 3 months post discharge from hospital
Population: Data were not collected from 2 participants from the Nicardipine arm and 5 participants in the Nicardipine + Verapamil + Nitroglycerin arm because the assessment was not administered to them.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicardipine | Verapamil | Nicardipine + Verapamil + Nitroglycerin
Number analyzed (Participants) | 30 | 30 | 24
score on a scale | 1.967 (1.771) | 1.759 (1.455) | 2.167 (2.140)

3. Other Pre Specified Outcome: Intra-cranial Pressure
Description: Intra-cranial pressure will be measured 1 day prior to vasospasm treatment and 1 day after vasospasm treatment
Time Frame: 1 day prior to procedure & 1 day after the procedure
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 3 months
Arm/Group | Nicardipine | Verapamil | Nicardipine + Verapamil + Nitroglycerin
All-Cause Mortality (participants affected / at risk) | 2/32 | 0/31 | 3/29
Serious Adverse Events (participants affected / at risk) | 4/32 | 0/31 | 5/29
Other Adverse Events (participants affected / at risk) | 21/32 | 13/31 | 27/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nicardipine (N=32) | Verapamil (N=31) | Nicardipine + Verapamil + Nitroglycerin (N=29)
Poor prognosis leading to death (General disorders) | 1 | 0 | 2
Subarachnoid hemorrhage leading to death (Nervous system disorders) | 1 | 0 | 0
respiratory failure secondary to Subarachnoid hemorrhage leading to death (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Elevated Intracranial Pressure (Nervous system disorders) | 0 | 0 | 1
Intracranial Hemorrhage (Nervous system disorders) | 1 | 0 | 0
Stroke (Nervous system disorders) | 0 | 0 | 1
recurrent subarachnoid hemorrhage (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicardipine (N=32) | Verapamil (N=31) | Nicardipine + Verapamil + Nitroglycerin (N=29)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Acute Posthemorrhagic Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 4 (4)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral Spinal Fluid Leak (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Dry Gangrene (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 1 (1) | 4 (4)
Elevated Intracranial Pressure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Fever (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 3 (3) | 6 (6) | 4 (4)
Hyponatremia (Renal and urinary disorders) | 3 (3) | 1 (1) | 3 (3)
Intracranial Hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Aysymptomatic NSTEMI (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Periorbital Edema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3)
Positive Culture (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pseudoaneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Subconjunctival Hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/36/NCT01996436/Prot_SAP_000.pdf